| Stay Connected: Testing an | Intervention to Comba | at COVID-19 Related | Social Isolation | Among Seattle- |
|---|---|---|---|---|
| | area Olo | der Adults | | |

NCT04966910

3/11/2021

**Statistical Analysis Plan.** We conducted Repeated Measure ANOVAs with time x condition interaction effects to facilitate statistical examination of rate of change over time for both conditions and impacts of condition on outcome. Sphericity tests were not significant for any model and is assumed in tests of within-subjects effects. Due to the small sample size and the lack of covariates associated with missing data, we were unable to conduct multiple imputation or other modeling approaches to missing data and therefore used a listwise missing approach. This provided 17 participants in the Stay Connected condition and 14 participants in the Usual Care condition.